CLINICAL TRIAL: NCT00219141
Title: A 36-week, Randomized, Double-blind, Multi-center, Parallel Group Study Comparing the Efficacy and Safety of Aliskiren in Combination With Losartan Compared to Losartan on the Regression of Left Ventricular Hypertrophy in Overweight Patients With Essential Hypertension
Brief Title: Aliskiren in Combination With Losartan Compared to Losartan on the Regression of Left Ventricular Hypertrophy in Overweight Patients With Essential Hypertension
Acronym: ALLAY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Novartis Pharmaceuticals, External Affairs
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2316
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Hypertension; Left Ventricular Hypertrophy; Overweight
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular; Overweight | interventions — aliskiren; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Aliskiren 300 mg (Experimental): Patients in this arm initially received 150 mg of aliskiren for two weeks and were then force-titrated up to 300 mg of aliskiren where they remained for 34 weeks. In order to adequately blind the study, patients were required to take a total of 2 tablets and 1 capsule of study medication or placebo per day. In the first 2 weeks, patients took 1 tablet of aliskiren 150 mg, 1 tablet of aliskiren 150 mg placebo, and 1 capsule of losartan placebo. In the remaining 34 weeks, patients took 2 tablets of aliskiren 150 mg and 1 capsule of losartan placebo. Each dose was to be taken by mouth with water at approximately 8:00 AM, except on the morning of study visit when the dose was taken after all procedures and assessments had been completed.
  Interventions: Drug: Aliskiren 150/300 mg; Drug: Aliskiren placebo; Drug: Losartan 50/100 mg placebo
- Losartan 100 mg (Active Comparator): Patients in this arm initially received 50 mg of losartan for two weeks and were then force-titrated up to 100 mg of losartan where they remained for 34 weeks. In order to adequately blind the study, patients were required to take a total of 2 tablets and 1 capsule of study medication or placebo per day. In the first 2 weeks, patients took 2 tablets of aliskiren 150 mg placebo and 1 capsule of losartan 50 mg. In the remaining 34 weeks, patients took 2 tablets of aliskiren 150 mg placebo and 1 capsule of losartan 100 mg. Each dose was to be taken by mouth with water at approximately 8:00 AM, except on the morning of study visit when the dose was taken after all procedures and assessments had been completed.
  Interventions: Drug: Losartan 50/100 mg; Drug: Aliskiren placebo
- Aliskiren/losartan 300/100 mg (Experimental): Patients in this arm initially received 150 mg of aliskiren in combination with 50 mg of losartan for two weeks and were then force-titrated up to 300 mg of aliskiren in combination with 100 mg of losartan where they remained for 34 weeks. In order to adequately blind the study, patients were required to take a total of 2 tablets and 1 capsule of study medication or placebo per day. In the first 2 weeks, patients took 1 tablet of aliskiren 150 mg, 1 tablet of aliskiren 150 mg placebo, and 1 capsule of losartan 50 mg. In the remaining 34 weeks, patients took 2 tablets of aliskiren 150 mg and 1 capsule of losartan 100 mg. Each dose was to be taken by mouth with water at approximately 8:00 AM, except on the morning of study visit when the dose was taken after all procedures and assessments had been completed.
  Interventions: Drug: Aliskiren 150/300 mg; Drug: Losartan 50/100 mg; Drug: Aliskiren placebo

INTERVENTIONS:
Drug: Aliskiren 150/300 mg — Aliskiren 150 mg tablets
  Arms: Aliskiren 300 mg; Aliskiren/losartan 300/100 mg
Drug: Losartan 50/100 mg — Losartan 50 or 100 mg capsules
  Arms: Aliskiren/losartan 300/100 mg; Losartan 100 mg
Drug: Aliskiren placebo — Aliskiren 150 mg placebo tablet
Drug: Losartan 50/100 mg placebo — Losartan 50/100 mg placebo capsules
  Arms: Aliskiren 300 mg

SUMMARY:
To compare the efficacy and safety of aliskiren in combination with losartan compared to losartan on the regression of the increased size of the left ventricle in overweight patients with high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential hypertension
* Patients with a BMI > 25 kg/m2
* Patients with LVH (LVWT ≥ 1.3 cm) confirmed by the ECHO

Exclusion Criteria:

* Patients treated with an ACE or an ARB within 3 months of study entry (Study Visit 1) who are unable or unwilling to undergo the 3 month washout period.
* Patients treated with an ACE and ARB combination at study entry.
* Known secondary hypertension of any etiology (e.g., uncorrected renal artery stenosis).

Other protocol related inclusion/exclusion criteria applied to the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2005-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- sites in Argentina, Argentina, Argentina
- sites in Colombia, Colombia, Colombia
- sites in Finland, Finland, Finland
- sites in Germany, Germany, Germany
- sites in Italy, Italy, Italy
- sites in Russia, Russia, Russia
- sites in Spain, Spain, Spain
- sites in Sweden, Sweden, Sweden

REFERENCES:
- [Derived] Wang GM, Li LJ, Fan L, Xu M, Tang WL, Wright JM. Renin inhibitors versus angiotensin receptor blockers for primary hypertension. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD012570. doi: 10.1002/14651858.CD012570.pub2. PMID 40013543
- [Derived] Pouleur AC, Uno H, Prescott MF, Desai A, Appelbaum E, Lukashevich V, Smith BA, Dahlof B, Solomon SD; ALLAY Investigators. Suppression of aldosterone mediates regression of left ventricular hypertrophy in patients with hypertension. J Renin Angiotensin Aldosterone Syst. 2011 Dec;12(4):483-90. doi: 10.1177/1470320311414453. Epub 2011 Jul 11. PMID 21746765

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren 300 mg: Patients in this arm initially received 150 mg of aliskiren for two weeks and were then force-titrated up to 300 mg of aliskiren where they remained for 34 weeks.
- Losartan 100 mg: Patients in this arm initially received 50 mg of losartan for two weeks and were then force-titrated up to 100 mg of losartan where they remained for 34 weeks.
- Aliskiren/Losartan 300/100 mg: Patients in this arm initially received 150 mg of aliskiren in combination with 50 mg of losartan for two weeks and were then force-titrated up to 300 mg of aliskiren in combination with 100 mg of losartan where they remained for 34 weeks.
Period: Overall Study
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Started | 154 | 152 | 154
Completed | 140 | 131 | 142
Not Completed | 14 | 21 | 12
Not completed — Adverse Event | 4 | 10 | 5
Not completed — Lack of Efficacy | 3 | 2 | 0
Not completed — Administrative problems | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 4 | 1
Not completed — Protocol Violation | 3 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 5
Not completed — Condition no longer requires study drug | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg | Total
Number analyzed (Participants) | 154 | 152 | 154 | 460
Age Continuous [Mean (Standard Deviation); unit: years] | 58.4 (9.61) | 59.2 (11.00) | 58.8 (10.62) | 58.8 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 35 | 35 | 112
  Male | 112 | 117 | 119 | 348

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular Mass Index (LVMI) From Baseline to End of Study (Week 36)
Description: Left ventricular mass index (LVMI) was measured by magnetic resonance imaging (MRI). An increase in LVMI indicates hypertrophy of the left ventricle. This could be a normal reversible response to cardiovascular conditioning (athletic heart) or an abnormal irreversible response to chronically increased volume load (preload) or increased pressure load (afterload). Thickening of the ventricular muscle results in increased left ventricular pressure, increased end-systolic volume, and decreased end-diastolic volume, causing an overall reduction in cardiac output.
Time Frame: Baseline to end of study (Week 36)
Population: Efficacy population: All patients who had a baseline measurement and at least one post-baseline efficacy variable measurement patients and who had been treated for at least 28 weeks and had evaluable MRI assessments both at baseline and at the end of the study.
Measure: Least Squares Mean (Standard Error); unit: g/m^2
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Number analyzed (Participants) | 132 | 123 | 136
g/m^2 | -5.51 (0.95) | -4.81 (0.98) | -5.61 (0.93)

2. Secondary Outcome: Change in the Left Ventricular Hypertrophy (LVH) Parameter Left Ventricular Mass Index as Measured by MRI From Baseline to End of Study (Week 36)
Time Frame: Baseline to end of study (Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Number analyzed (Participants) | 132 | 123 | 136
g/m^2 | -4.87 (11.69) | -4.79 (11.87) | -5.81 (10.93)

3. Secondary Outcome: Change in the Left Ventricular Hypertrophy (LVH) Parameter Left Ventricular End Diastolic Volume as Measured by MRI From Baseline to End of Study (Week 36)
Time Frame: Baseline to end of study (Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Number analyzed (Participants) | 132 | 123 | 134
mL | -7.05 (24.09) | -4.52 (25.15) | -7.03 (24.97)

4. Secondary Outcome: Change in the Left Ventricular Hypertrophy (LVH) Parameter Left Ventricular End Systolic Volume as Measured by MRI From Baseline to End of Study (Week 36)
Time Frame: Baseline to end of study (Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Number analyzed (Participants) | 132 | 123 | 134
mL | -3.20 (16.64) | -4.73 (15.16) | -5.14 (15.35)

5. Secondary Outcome: Change in the Left Ventricular Hypertrophy (LVH) Parameter Left Ventricular Anteroseptal Wall Thickness as Measured by MRI From Baseline to End of Study (Week 36)
Time Frame: Baseline to end of study (Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Number analyzed (Participants) | 132 | 123 | 134
mm | -0.95 (2.71) | -1.20 (2.56) | -1.17 (2.61)

6. Secondary Outcome: Change in the Left Ventricular Hypertrophy (LVH) Parameter Left Ventricular Inferolateral Wall Thickness as Measured by MRI From Baseline to End of Study (Week 36)
Time Frame: Baseline to end of study (Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Number analyzed (Participants) | 132 | 123 | 134
mm | -0.88 (2.03) | -0.89 (2.16) | -0.90 (2.22)

7. Secondary Outcome: Change in the Left Ventricular Hypertrophy (LVH) Parameter Diameter of Ascending Aorta as Measured by MRI From Baseline to End of Study (Week 36)
Time Frame: Baseline to end of study (Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Number analyzed (Participants) | 133 | 129 | 137
mm | -0.71 (1.72) | -0.64 (2.16) | -0.86 (2.06)

8. Secondary Outcome: Change in the Left Ventricular Hypertrophy (LVH) Parameter Left Ventricular End Diastolic Mass as Measured by MRI From Baseline to End of Study (Week 36)
Time Frame: Baseline to end of study (Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Number analyzed (Participants) | 132 | 123 | 134
g | -9.81 (23.84) | -9.92 (24.24) | -12.29 (22.58)

9. Secondary Outcome: Change in the Left Ventricular Hypertrophy (LVH) Parameter Left Ventricular Ejection Fraction as Measured by MRI From Baseline to End of Study (Week 36)
Time Frame: Baseline to end of study (Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Number analyzed (Participants) | 132 | 123 | 133
percent | 0.62 (7.73) | 2.02 (6.70) | 1.92 (7.00)

10. Secondary Outcome: Change in the Left Ventricular Hypertrophy (LVH) Parameter Left Ventricular Stroke Volume as Measured by MRI From Baseline to End of Study (Week 36)
Time Frame: Baseline to end of study (Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Number analyzed (Participants) | 132 | 123 | 133
mL | -3.89 (17.83) | 0.24 (17.53) | -2.24 (17.25)

11. Secondary Outcome: Change in the Left Ventricular Hypertrophy (LVH) Parameter Sokolow-Lyon Voltage as Measured by Electrocardiogram From Baseline to End of Study (Week 36)
Time Frame: Baseline to end of study (Week 36)
Population: Intent-to-treat population: All patients who had a baseline measurement and at least one post-baseline efficacy variable measurement.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Number analyzed (Participants) | 145 | 146 | 146
mm | -1.07 (3.78) | -0.97 (4.22) | -1.43 (3.81)

12. Secondary Outcome: Change in the Left Ventricular Hypertrophy (LVH) Parameter Cornell Voltage Duration Product as Measured by Electrocardiogram From Baseline to End of Study (Week 36)
Time Frame: Baseline to end of study (Week 36)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mm * ms
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Number analyzed (Participants) | 140 | 144 | 146
mm * ms | -104.97 (376.30) | -150.31 (439.81) | -130.65 (453.17)

13. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory Diastolic and Systolic Blood Pressure From Baseline to the End of the Study (Week 36)
Description: Two 24-hour ambulatory blood pressure monitoring (ABPM) evaluations were performed, one at baseline and one at the end of the study. For each evaluation, the ABPM device was attached to the non-dominant arm of the patient. A correlation was made between the ABPM device readings and measurements taken with a mercury sphygmomanometer and stethoscope. Following the correlation procedure, blood pressure was measured at study specified intervals.
Time Frame: Baseline the end of study (Week 36)
Population: Ambulatory blood pressure monitoring completers population: All patients that completed both ambulatory blood pressure monitoring assessments successfully.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Number analyzed (Participants) | 83 | 89 | 84
mm Hg
  Systolic | -2.67 (1.19) | -3.81 (1.17) | -6.97 (1.21)
  Diastolic | -1.31 (0.82) | -1.92 (0.81) | -4.11 (0.83)

ADVERSE EVENTS:
Arm/Group | Aliskiren 300 mg | Losartan 100 mg | Aliskiren/Losartan 300/100 mg
Serious Adverse Events (participants affected / at risk) | 10/154 | 13/152 | 10/154
Other Adverse Events (participants affected / at risk) | 31/154 | 31/152 | 29/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300 mg (N=154) | Losartan 100 mg (N=152) | Aliskiren/Losartan 300/100 mg (N=154)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Neuropathy (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300 mg (N=154) | Losartan 100 mg (N=152) | Aliskiren/Losartan 300/100 mg (N=154)
Diarrhoea (Gastrointestinal disorders) | 6 | 9 | 7
Nasopharyngitis (Infections and infestations) | 11 | 13 | 11
Dizziness (Nervous system disorders) | 5 | 3 | 8
Headache (Nervous system disorders) | 14 | 8 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.